CLINICAL TRIAL: NCT02104648
Title: A 2 PART STUDY IN HEALTHY SUBJECTS: PART A: A MULTIPLE DOSE, RANDOMIZED, PLACEBO CONTROLLED STUDY TO EVALUATE THE SAFETY AND TOLERABILITY OF SUPRA-THERAPEUTIC DOSES OF RO4602522; PART B: A MULTIPLE-DOSE, RANDOMIZED, DOUBLE-BLIND, DOUBLE DUMMY, PLACEBO CONTROLLED, POSITIVE-CONTROL, PARALLEL GROUP STUDY TO INVESTIGATE THE EFFECT OF RO4602522 ON THE QTC INTERVAL
Brief Title: A 2-Part Study to Evaluate the Safety of Supra-Therapeutic Doses of RO4602522 and to Investigate the Effect of RO4602522 on the QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP29269
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — sembragiline; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Part A: Placebo (Placebo Comparator)
  Interventions: Other: Placebo RO4602522
- Part A: RO4602522 (Experimental)
  Interventions: Drug: RO4602522
- Part B: RO4602522 Multiple Doses (Experimental)
  Interventions: Drug: RO4602522; Other: moxifloxacin placebo
- Part B: RO4602522 Single Dose (Experimental)
  Interventions: Other: Placebo RO4602522; Drug: RO4602522; Other: moxifloxacin placebo
- Part B: moxifloxacin Single Dose (Experimental)
  Interventions: Other: Placebo RO4602522; Drug: moxifloxacin

INTERVENTIONS:
Other: Placebo RO4602522 — Daily oral doses
  Arms: Part A: Placebo; Part B: RO4602522 Single Dose; Part B: moxifloxacin Single Dose
Drug: RO4602522 — Daily oral doses
  Arms: Part A: RO4602522; Part B: RO4602522 Multiple Doses
Drug: RO4602522 — Single, oral dose
  Arms: Part B: RO4602522 Single Dose
Drug: moxifloxacin — 400 mg oral dose given on Day 1 or 11
  Arms: Part B: moxifloxacin Single Dose
Other: moxifloxacin placebo — Dose given orally on Days 1 and/or 11
  Arms: Part B: RO4602522 Multiple Doses; Part B: RO4602522 Single Dose

SUMMARY:
This is a 2 part study to evaluate the safety and tolerability of supra-therapeutic doses of RO4602522 (Part A); and to investigate the effect of RO4602522 on the QTcF interval in healthy volunteers (Part B). Part A of the study will be a multiple-dose, randomized, double-blind, placebo-controlled study. Participants will be randomized to receive daily, oral doses of either RO4602522 or placebo for ten days. Part B of the study will be a multiple-dose, randomized, double-blind, double-dummy, placebo controlled, positive-control, parallel group study. Participants will be randomized to receive either multiple or single doses of RO4602522 or to receive single doses of moxifloxacin for 11 days. Pharmacokinetic parameters will be assessed for Parts A and B; and continuous ECG recordings will be made during Part B.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 65 years of age, inclusive. For Part B: Healthy male and female subjects, 18 to 65 years of age, inclusive (female subjects only if the repeat dose is tolerated in Part A)
* Healthy status is defined by absence of evidence of any clinically significant, active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology and urinalysis
* A BMI between 18 to 32 kg/m2 inclusive
* Use of highly effective contraception

Exclusion Criteria:

* Pregnant or breast-feeding women
* Suspicion of alcohol or drug abuse or positive drug screen
* Positive result on hepatitis B (HBsAg), hepatitis C (HCV), or HIV 1 and 2
* History of any clinically significant gastrointestinal, renal, hepatic, broncho-pulmonary, neurological, psychiatric, cardio-vascular, endocrinological, hematological or allergic disease, metabolic disorder, cancer or cirrhosis
* Diseases or medical conditions that are capable of altering the absorption, metabolism or elimination of drugs
* Any prescribed or over-the-counter medications (including vitamins or herbal remedies) taken within 2 weeks prior to first dosing or within 5 times the elimination half-life of the medication prior to first dosing (whichever is longer)
* Taking any nutrients known to modulate CYP3A activity (e.g., grapefruit juice; Seville orange) within 2 weeks prior to administration of study drugs or tyramine rich nutrients 48 hours prior to admission to study site and then throughout the study
* Participation in an investigational drug or device study within 60 days prior to screening or 5 times the elimination half-life of the medication prior to first dosing (whichever is longer)
* Consumption of nicotine and/ or tobacco products within the last 45 days prior to Day 1 of study

Part B

* Any clinically significant cardiovascular findings or history of such
* Allergy to moxifloxacin or any quinolone antibiotics or history of tendon rupture with quinolone-type antibiotic or any confirmed clinically significant allergic reactions against any drug, or multiple allergies in the judgment of the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Part A: Incidence of adverse events | Up to 30 days
Part B: Continuous, 12-lead, Holter electrocardiogram (ECG) recordings | Days -1 (screening) to 11

SECONDARY OUTCOMES:
Parts A & B: Area under the concentration-time curve (AUC) of RO4602522 | Days 1 to 10

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Lenexa, Kansas, United States